CLINICAL TRIAL: NCT00997490
Title: Phase III Placebo-controlled, Randomised, Single-centre, Double-blind Study of the Antidepressant Efficacy of a Combination Herbal Drug Preparation
Brief Title: Study of the Antidepressant Efficacy of a Combination Herbal Drug Preparation (NEURAPAS Balance)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Clearly identifiable benefits 50% of patients included
Sponsor: Pascoe Pharmazeutische Praeparate GmbH (Industry)
Responsible Party: Anja Braschoss, Pascoe Pharmazeutische Preparate GmbH
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSC 120/99
Record Dates: First submitted 2009-10-16; First posted 2009-10-19 (Estimated); Last update posted 2010-05-17 (Estimated); Status verified 2010-05

CONDITIONS: Depressive Disorder
Keywords: depression; HAMD 21; anxiety; HAMA; Hypericum; Valerian; Passionflower; F32.0; F33.0
MeSH Terms: conditions — Depressive Disorder; Depression; Anxiety Disorders | interventions — Valeriana extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Verum (Experimental): Neurapas balance, film-coated tablet
  Interventions: Drug: Neurapas® balance (Herbal combination out of hypericum, valerian, passionflower)
- Placebo (Placebo Comparator)
  Interventions: Drug: film-coated sugar-pill

INTERVENTIONS:
Drug: Neurapas® balance (Herbal combination out of hypericum, valerian, passionflower) — 3 x 2 tablets/day over 6 weeks
  Other Names: Neurapas balance, film-coated tablet
  Arms: Verum
Drug: film-coated sugar-pill — 3 x 2 tablets / day over 6 weeks
  Arms: Placebo

SUMMARY:
The efficacy and tolerability of Neurapas® balance was compared against placebo in this single-centre, controlled, double-blind study in patients with a mild depressive episode.

After a one-week placebo run-in phase to exclude placebo responders, patients were given the study medication (Neurapas® balance or placebo) for 6 weeks in a dose of 3 x 2 tablets daily.

The improvement in symptoms of depression was assessed on the basis of the internationally established Hamilton Depression Scale 21. The Self-Rating Depression Scale (SDS), the Hamilton Anxiety Scale (HAM-A), the Clinical Global Impressions (CGI), Quality of Life questionnaire (SF-36) according to Bullinger (German version) and a Sleep questionnaire (SQ) were used as further efficacy criteria.

DETAILED DESCRIPTION:
The efficacy and tolerability of Neurapas® balance was compared against placebo in this single-centre, controlled, double-blind study in patients with a mild depressive episode according to ICD 10, F32.0 and F33.0.

After a one-week, placebo run-in phase to exclude placebo responders, patients were given the study medication (Neurapas® balance or placebo) for 6 weeks in a dose of 3 x 2 tablets daily. The study was conducted in accordance with the relevant requirements of the German Medicines Act (AMG), the Declaration of Helsinki (48th General Assembly, Sommerset West, Rep. of South Africa, October 1996) and ICH GCP guidelines.

The improvement in symptoms of depression was assessed on the basis of the internationally established Hamilton Depression Scale 21 (primary efficacy criterion). The Self-Rating Depression Scale (SDS), the Hamilton Anxiety Scale (HAM-A), the Clinical Global Impressions (CGI), Quality of Life questionnaire (SF-36) according to Bullinger (German version) and a Sleep questionnaire (SQ) were used as secondary efficacy criteria.

ELIGIBILITY:
Inclusion Criteria:

* Depressive symptoms of mild intensity, as defined in the International Classification of Mental Disorders (ICD 10), codes F32.0 (mild depressive episode) and F33.0 (recurrent depressive disorder, current episode mild)
* SDS Index between 51 and 59 (this criterion was declared null and void on 21.02.02 in the 2nd Amendment)
* HAM-D21 scores between 10 and 17
* Between 18 and 70 years of age
* Duration of depression: not less than 4 weeks and not longer than 2 years
* Signed informed consent to take part in the clinical study after verbal and written information.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2001-01; Primary Completion 2002-07 (Actual); Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
HAM-D 21 | Visit 1 (Start of medication), Visit 2 (End of run-in phase), Visit 4 (after 2 weeks treatment), Visit 6 (after 4 weeks treatment), Visit 8 (End of Study)

SECONDARY OUTCOMES:
Self-Rating Depression Scale (SDS) | V1, V2, V4, V6, V8
HAMILTON Anxiety Scale (HAM-A) | V2, V4, V6, V8
Clinical Global Impressions (CGI) | V2, V8
BULLINGER Quality of Life questionnaire (SF-36) | V2, V6, V8
Sleep questionnaire (SQ) | V2, V6, V8

CONTACTS AND LOCATIONS:
Overall Officials: Ilie Urlea-Schoen, Dr med (RO), Principal Investigator; Anja Braschoss, MD, Study Director — Pascoe Pharmazeutische Praeparate GmbH
Locations (1):
- Dr. Urlea-Schoen, Siegen, North Rhine-Westphalia, Germany